CLINICAL TRIAL: NCT04944485
Title: One Year Clinical Performance of Self Adhesive Giomer Containing Flowable Composite in Restoring Class V Cavities: A Randomized Clinical Trial
Brief Title: One Year Clinical Performance of Self Adhesive Giomer Containing Flowable Composite in Restoring Class V Cavities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Salma Mohamed Monir Mahmoud Ahmed, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14422019423506
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Class V Dental Caries; Composite Resin and Self Adhesive Flowable Composite
MeSH Terms: interventions — CMW cement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The assessors, statistician and the patients will be blinded to intervention/control assessment methods; Triple blinded study. Also, it will not be allowed amongst the examiners to exchange any information throughout the entire study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- class V cavities treated with putty nanohybrid resin composite (Active Comparator): Selective enamel etching will be done and a universal adhesive (Prime&Bond universal™ ,Dentsply)will be applied to both enamel and dentin. After gentle dryness and solvent evaporation the bonding agent will be cured for 20 seconds. Composite (Neo Spectra™ST, Dentsply, Sirona, USA) will be placed incrementally and light cured for 20 seconds
  Interventions: Other: (Neo Spectra™ ST, Dentsply, Sirona, USA)
- class V cavities treated with Self adhesive giomer containing nanohybrid flowable composite (Experimental): Cleaning and gentle air blowing of the preparation. Then applying FIT SA F03 (Low Flow), SHOFU, USA. Spread in a thin layer (≤0.5mm) on the prepared surface with needle tip, microbrush and gently air-blow leave for 20 seconds then light cure for 5 seconds. Then,apply additional increments (≤2mm) of FIT SA and light cure each increment for 10 seconds then finish and polish
  Interventions: Other: (FIT SA F03, SHOFU, USA)

INTERVENTIONS:
Other: (FIT SA F03, SHOFU, USA) — Self adhesive giomer containing nanohybrid flowable composite
  Arms: class V cavities treated with Self adhesive giomer containing nanohybrid flowable composite
Other: (Neo Spectra™ ST, Dentsply, Sirona, USA) — Conventional technique using putty nanohybrid resin composite
  Arms: class V cavities treated with putty nanohybrid resin composite

SUMMARY:
This clinical trial will be conducted to compare the clinical performance of self adhesive giomer containing flowable composite and putty nanohybrid resin composite in class V cavities over one year follow-up

DETAILED DESCRIPTION:
This clinical trial will be conducted in Department of Conservative Dentistry, Faculty of Dentistry,Cairo university outpatient clinic. The Operator in charge will be: Salma Mohamed Monir (S.M).

The researcher will bear ultimate responsibility for all activities associated with the conduct of a research project including recruitment of patients, explaining and performing the procedures to the patients.

Screening of patients that come to the Conservative Dentistry Department Clinic seeking dental care will continue until the target population is achieved. The patients will be subjected to full examination and diagnosis using dental charts. Once the patients that are potentially eligible for this study are identified, the patients will be contacted by the research investigator (S.M) who will explain the study and ascertains the patient's interest. If interested, more detailed evaluations and preparations are made.

Randomization will be done using simple randomization by (N.K) by generating numbers from 1:100 into two columns according to interventions/Control assessment methods. The allocation sequence will be generated using (www.randomization.com) The randomization list will be kept with (N.K) and will be kept secured away to ensure no tampering with the random list. Each participant will choose a random number from an opaque sealed envelope. When the participant chooses an envelope, it will be signed by the patient and the supervisor and the number on the envelope will be recorded in the patient chart to ensure that the patient is assigned to the randomized group The assessors, statistician and the patients will be blinded to intervention/control assessment methods; Triple blinded study. Also, it will not be allowed amongst the examiners to exchange any information throughout the entire study period.

For every patient medical and dental history will be taken. Examination charts will be filled by the investigator S.M.

Informed consent:

Patients attending at the Department of Conservative Dentistry, Faculty of Dentistry, Cairo University will be screened. Those who meet the study inclusion criteria will be recruited, will be informed with the study and an informed consent will be signed if the patients approve.

Periodontal treatment:

Periodontal treatment will be made and oral hygiene instructions will be enforced. Then, the operator will start rubber-dam isolation and cavity preparation is done as follows:

Cavity preparation procedure:

Patients will be given local anesthesia as required, and the teeth will be isolated. A No. #330 bur (0.8 mm in diameter and 1.6 mm in length) in a high speed hand piece with air /water coolant will be used to prepare class V cavity preparations. Any tooth that will suffer from pulpal exposure will be excluded from the study. Remaining caries will be excavated by a sharp excavator. A 1mm bevel will be prepared in enamel margins (Folwaczny et al., 2001). According to the concealed envelope, the tooth will be assigned to one of both treatment groups.

Control group: Selective enamel etching will be done and a universal adhesive (Prime&Bond universal™ ,Dentsply)will be applied to both enamel and dentin. After gentle dryness and solvent evaporation the bonding agent will be cured for 20 seconds. Composite (Neo Spectra™ST, Dentsply, Sirona, USA) will be placed incrementally and light cured for 20 seconds (Noé Orellana et al., 2009)

Intervention group: Cleaning and gentle air blowing of the preparation. Then applying FIT SA F03 (Low Flow), SHOFU, USA. Spread in a thin layer (≤0.5mm) on the prepared surface with needle tip, microbrush and gently air-blow leave for 20 seconds then light cure for 5 seconds. Then, apply additional increments (≤2mm) of FIT SA and light cure each increment for 10 seconds then finish and polish.

Post curing will be done using glycerin to decrease the oxygen inhibited layer (Strnad et al.,2015). Finishing will be done using yellow and white finishing stones. More finishing and polishing will be done. Rubber-dam will be removed and patients will be recalled for evaluation after 3, 6 and 12 months. A.R and Y.S will be blinded to both treatment groups. AR and Y.S will give the restorations a score using Modified USPHS score.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with carious anterior or posterior buccal class V lesions.
2. No signs of irreversible pulpitis (vital teeth)
3. Young adult males or females.
4. . Acceptable oral hygiene.
5. Co-operative patients approving to participate in the study

Exclusion Criteria:

1. Patients with a compromised medical history.
2. Severe or active periodontal disease
3. Systemic diseases or severe medical complications (disabilities).
4. Lack of compliance
5. Extensive carious lesion that is in risk of pulp exposure.
6. Rampant caries.
7. History of pain or swelling.
8. Endodontically treated teeth.
9. Mobility grade 1 or 2
10. Non-carious cervical abfraction lesions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Assessing change in marginal discoloration between time points 3, 6 ,12 months | 3,6,12 months
  Visual inspection with mirror Alpha :There is no visual evidence of any marginal discoloration at the junction of the restoration and the adjacent tooth structure . Bravo :There is visual evidence of shallow marginal discoloration. Charlie : There is visual evidence of deep marginal discoloration toward a pulpal direction.

SECONDARY OUTCOMES:
Assessing change in modified USPHS criteria between time points 3, 6 ,12 months | 3,6,12 months
  visual inspection of postoperative hypersensitivity ,secondary caries, gross fracture,colour match , marginal integrity , anatomic contour and surface texture

IPD SHARING:
Plan to Share IPD: No